CLINICAL TRIAL: NCT00751218
Title: A Comparative Double-Blind, Double- Dummy Study of Desloratadine (DL) 5 MG Once Daily, Cetirizine 10 MG Once Daily, and Placebo Once Daily in Patients With Chronic Idiopathic Urticaria (CIU)
Brief Title: A Comparative Double-Blind, Double- Dummy Study of Desloratadine (DL) 5 MG Once Daily, Cetirizine 10 MG Once Daily, and Placebo Once Daily in Patients With Chronic Idiopathic Urticaria (Study P03735)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P03735
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Urticaria
MeSH Terms: conditions — Urticaria | interventions — desloratadine; Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Active Comparator): desloratadine
  Interventions: Drug: desloratadine
- Arm 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- Arm 3 (Active Comparator): cetirizine
  Interventions: Drug: cetirizine

INTERVENTIONS:
Drug: desloratadine — desloratadine, 5mg oral tablets, once daily for 28 days
  Other Names: SCH 034117
  Arms: Arm 1
Drug: placebo — placebo, once daily for 28 days
  Arms: Arm 2
Drug: cetirizine — cetirizine, 10 mg capsules once daily for 28 days
  Arms: Arm 3

SUMMARY:
This was a randomized, double-blind, parallel-group, multicenter study that used both an active control (cetirizine) and a placebo control to evaluate desloratadine 5 mg once daily during a 28-day treatment period. The active treatments and placebo were allocated in a 2:2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Have demonstrated their willingness to participate in the study and comply with its procedures by signing a written informed consent. For pediatric patients, the parent or legal guardian was to have signed a written informed consent.
* Be between 12 and 70 years of age, of either sex and any race.
* Had signs and symptoms of CIU for at least 6 weeks prior to the Screening Visit.
* Have been experiencing a current flare of their CIU of at least 3 weeks prior to the Baseline Visit. Hives were to have been present for at least 3 days per week during the current flare prior to the Baseline Visit.
* Have an overall condition of CIU that was at least of "moderate" severity (minimum score of 2) at both Screening and Baseline Visits.
* Have at least a moderately severe pruritus score (minimum score of 2) and hives (minimum score of 1) present at Screening.
* Have, at Baseline, a total pruritus score of >= 14 for the sum of AM and PM (reflective) diary scores for the 3 days prior to Baseline and the AM diary score on Day 1.
* Understand and be able to adhere to the dosing and visit schedules, and agree to assess and record their symptom severity scores, medication times, concomitant medications, and adverse events accurately and consistently in a daily diary.
* Be in general good health and free of any clinically significant disease (other than CIU) that would have interfered with study evaluations.
* If female and of childbearing potential, have had a negative urine (hCG) pregnancy test at the time of Baseline (Visit 2).
* Female subjects of childbearing potential were to be counseled in the appropriate use of birth control while in the study. They were to be using a medically accepted method of birth control

Exclusion Criteria:

* Had asthma requiring chronic use of inhaled or systemic corticosteroids.
* Had been unresponsive to antihistamine treatment in the past.
* Had a history of allergies to more than two classes of medication or who were allergic to or unable to tolerate antihistamines.
* Had used any investigational drug in the last 30 days prior to Baseline.
* Had food or drug allergies manifested as skin reactions. Subjects with urticaria that was primarily due to physical urticaria or other known etiology.
* If female, were pregnant or nursing.
* Had a history of hypersensitivity to the study drug or its excipients.
* Were family members of the investigational study staff involved with this study.
* Had previously been randomized into the study.
* Had current evidence of clinically significant hematopoietic, cardiovascular, hepatic, renal, neurologic, psychiatric, autoimmune disease, or other disease that precluded the subject's participation in the study. Particular attention was to be given to subjects with conditions that would interfere with the absorption, distribution, metabolism, or excretion of the study medication or with the subject's ability to reliably complete the diary card.
* Were morbidly obese (BMI >= 35, as described in Appendix 6 of the protocol)
* Had a compromised ability to provide informed consent.
* Had a history of non-compliance with medications or treatment protocols.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2004-05-06 (Actual); Primary Completion 2005-05-24 (Actual); Study Completion 2005-05-24 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy of the study treatments with respect to the change from Baseline in the average AM/PM 12-hour reflective pruritus severity score (diary recordings) after the first 7 days of treatment. | 7 days

SECONDARY OUTCOMES:
Joint physician-patient evaluations ("now") at treatment days 14 and 28 (Visit 3 and 4) of overall condition of the CIU and overall global therapeutic response | Days 14 and 28 (visits 3 and 4)
Average AM/PM "reflective" diary scores over for: severity of pruritus; number of hives; size of largest hives; total symptom score; subject-evaluated CIU interference with sleep (AM) and interference with daily activities (PM). | Treatment days 1-7, 8-14, 15-21 and 22-28
Adverse event reports and vital sign evaluations | Upon occurance